CLINICAL TRIAL: NCT06999915
Title: Influence of Individual Phenotypical Dimension (IPD) on Hard Tissue Stability Following Lateral Bone Augmentation: a Two-centre Clinical Study
Brief Title: The Effect of IPD on Lateral Bone Augmentation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRAS Project ID: 358068
Record Dates: First submitted 2025-05-09; First posted 2025-05-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Guided Bone Regeneration; Bone Resorption; Diagnostic Imaging
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the intervention, clinicians performing the surgical intervention and primary outcome examiner will be unblinded. Conversely, participants and researchers analyzing secondary outcomes (e.g., intra-oral & extra-oral scans, aesthetic scores) will be blinded to treatment allocation throughout the whole study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Test Group): IP and GBR as an over-contour augmentation beyond IPD (Experimental): Implant placement and simultaneous guided bone regeneration (GBR) beyond Individual Phenotypical Dimension (IPD). In this group, lateral bone augmentation will be performed as an over-contour augmentation of 3 mm beyond IPD.
  Interventions: Procedure: Group 1 (Test Group): IP and GBR as an over-contour augmentation beyond IPD
- Group 2 (Control Group): IP and GBR as a contour augmentation up to IPD (Active Comparator): Implant placement and simultaneous guided bone regeneration (GBR) up to IPD. In this group, lateral bone augmentation will be performed up to IPD
  Interventions: Procedure: Group 2 (Control Group): IP and GBR as a contour augmentation up to IPD

INTERVENTIONS:
Procedure: Group 1 (Test Group): IP and GBR as an over-contour augmentation beyond IPD — In this group, a bone level implant (Straumann BLC, SLActive®, Roxolid, Straumann AG, Switzerland) will be placed in an ideal 3D prosthetically guided position to allow for a screw-retained restoration, following the manufacturer's protocol. Guided bone regeneration (GBR) will be performed simultaneously with the implant placement with the aim to re-establish the original bone contour as defined by IPD. A bovine bone mineral graft (Bio-Oss collagen®, Geistlich, Wolhusen, Switzerland) will be placed on the buccal aspect of the implant and covered with a collagen membrane (Bio-Gide®, Geistlich, Wolhusen). In the test group, bone augmentation will be performed by adding biomaterial 3 mm beyond the Individual Phenotypical Dimension (IPD) to achieve over-contour augmentation. IPD will be clinically defined during surgery by connecting the most labially prominent points of adjacent ridges at the level of the bone zenith of neighboring teeth.
  Arms: Group 1 (Test Group): IP and GBR as an over-contour augmentation beyond IPD
Procedure: Group 2 (Control Group): IP and GBR as a contour augmentation up to IPD — In this group, a bone level implant (Straumann BLC, SLActive®, Roxolid, Straumann AG, Switzerland) will be placed in an ideal 3D prosthetically guided position to allow for a screw-retained restoration, following the manufacturer's protocol. Guided bone regeneration (GBR) will be performed simultaneously with the implant placement with the aim to re-establish the original bone contour as defined by IPD. A bovine bone mineral graft (Bio-Oss collagen®, Geistlich, Wolhusen, Switzerland) will be placed on the buccal aspect of the implant and covered with a collagen membrane (Bio-Gide®, Geistlich, Wolhusen). In the control group, bone augmentation will be performed by adding biomaterial up to the IPD line in order to achieve a contour augmentation with bone grafting remaining within the boundaries defined by the IPD. IPD will be clinically defined during surgery by connecting the most labially prominent points of adjacent ridges at the level of the bone zenith of neighboring teeth
  Arms: Group 2 (Control Group): IP and GBR as a contour augmentation up to IPD

SUMMARY:
Guided Bone Regeneration (GBR) is a widely used technique during dental implant surgery to help rebuild bone around the implant and improve its long-term appearance and stability. This study investigates whether the amount of bone that regrows depends on a person's original bone shape, known as the Individual Phenotypical Dimension (IPD). The aim is to compare the bone stability and overall results between two approaches: adding bone only up to the original bone line (IPD) or adding bone beyond it (over-contour augmentation). Over the course of a year, the study will assess not only bone and soft tissue healing, but also gum blood flow, implant success, and patient satisfaction.

There will be two treatment groups in this study - one group will receive bone grafting just up to their natural bone shape, while the other group will receive a slightly larger graft that extends about 3 mm beyond it. Throughout the study CBCT scans will be taken to assess bone changes around the implant area in order to measure how the bone shape and thickness change over time after surgery.

DETAILED DESCRIPTION:
This is a two-centre, prospective, non-inferiority clinical trial with two parallel study groups aimed at radiographically comparing the differences in hard tissue (lateral augmentation) stability following different GBR treatment protocols (contour augmentation or over-contour augmentation). The study consists of 12 visits over a period of approximately 16 to 18 months.

The study will take place at the Centre for Oral Clinical Research (COCR), at the Institute of Dentistry, Faculty of Medicine and Dentistry, Queen Mary University of London under The Royal London Dental Hospital, Barts Health NHS Trust, United Kingdom (leading centre) and at Implant Research Centre & Department of Periodontology, School of Dental Medicine, University of Belgrade, Serbia, according to local guidelines and procedures/interventions detailed below.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) patients
* Good medical and psychological health
* Engaged patients presenting with a Full Mouth Plaque Score (FMPS) of ≤ 20% within the 6 weeks prior to enrolment
* Need of a tooth/teeth replacement in the incisor, canine or premolar maxillary region that could be provided with an implant-supported fixed prosthesis
* A relatively symmetrical maxillary arch
* A nearly intact contra-lateral alveolar ridge
* At least one neighbouring natural tooth present with healthy periodontal conditions
* After implant placement, presence of a buccal bone dehiscence/ fenestration or buccal bone plate thickness of ≤ 1.5 mm requiring GBR (Monje et al., 2022; Jensen et al.,2023, Group 1 ITI Consensus Report).
* At least 4 weeks of post-extraction socket healing and no ridge preservation prior to implant placement.
* No acute infection at the site; adequate availability of bone apical and palatal to obtain implant primary stability
* A functional occlusion with a minimum of 4 occlusal units (i.e., pairs of occluding posterior teeth)
* Willingness to read and sign a copy of the Informed Consent Form (ICF) after reading the Patient Information Sheet (PIS), and after the nature of the study has been fully explained and potential questions fully answered.

Exclusion Criteria:

* Any known systemic disease severely affecting bone metabolism (e.g., Cushing's syndrome, Crohn's disease, rheumatoid arthritis, osteoporosis or diabetes type I and uncontrolled diabetes type II).
* Self-reported HIV or other severe immunosuppression.
* Self-reported alcoholism or chronic drug abuse.
* Heavy smokers ( > 10 cigarettes/day)
* Patients reporting use of vape/e-cigarettes
* Self-reported pregnancy or lactation
* Chronic treatment (i.e., 2 weeks or more) with any medication known to affect oral status or bone metabolism (e.g., bisphosphonates, hormone replacement therapy, immunosuppressants) within 1 month before baseline visit.
* Chronic treatment with anticoagulants (including Aspirin), corticosteroids, immunosuppressants or other medications that may influence blood coagulation/count.
* Untreated caries lesions in neighbouring teeth and untreated/uncontrolled periodontal disease; If patients require periodontal treatment (non-surgical and/or surgical), this will be arranged outside the study protocol and completed prior to enrolment;
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene in the area of implant placement.
* Patients requiring maxillary sinus lift surgery before implant placement or presenting bone dimensions (at any time point of the study) that do not allow implant placement or there is no clinical indication to perform study procedures (i.e. bone augmentation, implant placement).
* Patients not willing to receive animal-derived biomaterials for GBR.
* Patients suffering from a known psychological disorder or with limited mental capacity or language skills such that study information could not be understood, informed consent could not be obtained, or simple instructions could not be followed.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Linear dimensional (LD) changes of the buccal aspect of the augmented alveolar ridge | baseline, immediately after implant placement (IP) and 12 months after implant loading (IL)
  The primary objective is to compare radiographically the differences in the hard tissue stability (linear dimensional changes of the augmented ridge) following guided bone regeneration (GBR) simultaneous to implant placement (IP), when lateral bone augmentation is performed up to Individual Phenotypical Dimension (IPD) (control group) or as an over-contour augmentation beyond IPD (test group).

SECONDARY OUTCOMES:
Cross-sectional area changes of the buccal aspect of the augmented ridge | baseline, immediately after IP and 12 months after IL
  Cross-sectional area changes of the buccal aspect of the augmented ridge across the whole length of the implant (mm) (ROI) from the time of implant placement (IP) to 12 months after implant loading (IL), assessed by superimposing and comparing CBCT data from different visits.
Blood flow changes | baseline, immediately after, and at 1, 3, 7, 15, 30 days after IP
  Blood flow changes at baseline, immediately after, and at 1, 3, 7, 15, 30 days after IP
Soft tissue volume changes | baseline, immediately after, and at 1, 3, 7, 15, 30 days after IP, immediately after IL, 6 and 12 months after IL
  Soft tissue volume changes at baseline, immediately after, and at 1, 3, 7, 15, 30 days after IP, immediately after IL, 6 and 12 months after IL
Extra-oral 3D geometric changes | baseline, immediately after, 1, 3, 7, 15 and 30 days after IP
  Extra-oral 3D geometric changes assessed with a facial chairside scanner at baseline, immediately after, 1, 3, 7, 15 and 30 days after IP
Full mouth plaque score (FMPS) | baseline, 6 and 12 months after IL
  FMPS will be recorded as a percentage of total surfaces (6 sites per tooth/implant), which reveal the presence of plaque. A binary score will be assigned to each surface (1 for plaque present, 0 for absent).
Full mouth bleeding score (FMBS) | baseline, 6 and 12 months after IL
  FMBS will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of bleeding within 10 - 30 seconds following periodontal probing. A binary score will be assigned to each surface (1 for bleeding present, 0 for bleeding absent).
Probing pocket depth (PPD) | baseline, 6 and 12 months after IL
  PPD will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/ implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual)
Gingival recession (REC) | baseline, 6 and 12 months after IL
  REC will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/ implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual)
Clinical attachment level (CAL) | baseline, 6 and 12 months after IL
  CAL will be calculated considering the values for PPD and REC in mm
Suppuration | baseline, 6 and 12 months after IL
  Suppuration will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of suppuration following periodontal probing. A binary score will be assigned to each surface (1 for suppuration present, 0 for suppuration absent)
Implant success/survival | 6 and 12 months after IL
  Implant success will be based on well-defined criteria by Albrektsson et al. (1986) and survival defined as any dental implant which remained in situ (ITI consensus 2004) 6 and 12 months after IL. Modified success criteria will be applied to incorporate the aesthetic outcomes in success rates
Changes in the pink esthetic score (PES) | immediately after IL, 6 and 12 months after IL
  Changes in the pink esthetic score (PES) from loading to 6 and 12 months after loading.
  PES is a cumulative score, where seven variables are evaluated using a 0-1-2 scoring system, with the scores 14 and 0 being the best and the worst outcomes, respectively
Changes in the white esthetic score (WES) | immediately after IL, 6 and 12 months after IL
  Changes in the white esthetic score (WES) from loading to 6 and 12 months after loading.
  The WES is a cumulative score where five subgroups are assessed using a 0-1-2 scoring system, with the scores 10 and 0 being the best and the worst outcomes, respectively
Early healing index | 1, 3, 7, 15 days after IP
  Visual assessment of gingival healing and recording of wound healing (Wachtel et al., 2003) will be assessed during follow-ups at 1, 3, 7 and 15 days after the surgical intervention.
Patient satisfaction | immediately after IL, 6 and 12 after IL
  Each patient will be asked to rate their functional and aesthetic satisfaction regarding the overall implant treatment using a subjective outcome questionnaire immediately after IL, 6 and 12 after IL. The questionnaire includes seven questions to be answered in a 5-level Likert scale (poor; fair; good; very good; excellent) (Fava, Lin, Zahran, & Jokstad, 2015).
Life impact questionnaire | 1, 3, 7 and 15 days after IP
  Numerical rating scale (NRS) ranging from 0-10 will be complemented with a questionnaire to assess post-surgical pain and swelling at 1, 3, 7 and 15 days.
Patients' aesthetic satisfaction | immediately after IL, 6 and 12 months after IL
  A visual analogue scale (VAS) rating the overall patients' aesthetic perception of final restoration will also be recorded on the day of the implant loading with monolithic zirconia screw-retained crowns to 6 and 12 months after IL (Aitken, 1969). The scale will range from 0 (very poor aesthetics) to 10 (excellent aesthetics) and the subject can indicate the degree of satisfaction by marking vertically across the VAS scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Mardas, DDS, MS, PhD, Principal Investigator — QMUL
Locations (1):
- Barts Health NHS Trust Dental Hospital, London, United Kingdom